CLINICAL TRIAL: NCT01721564
Title: Pulmonary Artery Remodelling With Bosentan
Brief Title: Bosentan and Pulmonary Endothelial Function
Acronym: PARBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof David S Celermajer (Other)
Responsible Party: Sponsor-Investigator, Prof David S Celermajer, Scandrett Professor of Cardiology, Royal Prince Alfred Hospital, Sydney, Australia
Organization: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05-0255
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan

ARMS (1):
- Bosentan (Experimental): 62.5 mg Bosentan twice a day for 1 month 125 mg Bosentan twice a day for 5 months
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — 62.5 mg Bosentan twice a day for 1 month 125 mg Bosentan twice a day for 5 months

SUMMARY:
6 months therapy of Bosentan, an endothelin antagonist, will lead to improvement in pulmonary microvascular endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary arterial hypertension; idiopathic and connective tissue disease associated
* Confirmed or invasive haemodynamic:
* Mean pulmonary arterial pressure greater than or equal to 25 millimeters of mercury
* Pulmonary capillary wedge pressure less than 15 millimeters of mercury
* No prior pulmonary hypertension specific therapy
* Ability to provide informed consent

Exclusion Criteria:

* Contra-indications to medications used to test endothelial function; acetylcholine, sodium nitroprusside, NG-Monomethyl-L-Arginine, L-arginine
* Advanced renal disease
* Previous allergic reaction to contrast agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Celermajer, MBBS, PhD, DSc, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bosentan
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bosentan: 62.5 mg Bosentan b.i.d. for 1 month 125 mg Bosentan b.i.d. for 5 months
Arm/Group | Bosentan
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  Australia | 8

OUTCOME MEASURES:

1. Primary Outcome: Acetylcholine Vascular Reactivity Response
Description: Percent pulmonary flow change from baseline after acetylcholine
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Bosentan
Number analyzed (Participants) | 8
percentage of baseline | 180 (20)

2. Secondary Outcome: Intravascular Ultrasound - Pulmonary Artery Wall Thickness
Description: Change in intima-media thickness
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Bosentan
Number analyzed (Participants) | 8
percentage of baseline | 34 (2)

ADVERSE EVENTS:
Arm/Group | Bosentan
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes